CLINICAL TRIAL: NCT02674217
Title: Outpatient Hematopoietic Grafting in Patients With Multiple Sclerosis Employing Autologous Non-cryopreserved Peripheral Blood Stem Cells: A Feasibility Study
Brief Title: Outpatient Hematopoietic Grafting in Multiple Sclerosis Employing Autologous Peripheral Blood Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro de Hematología y Medicina Interna (Other)
Responsible Party: Principal Investigator, Guillermo J. RUIZ-ARGÜELLES, Director, Centro de Hematología y Medicina Interna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CentroHMI; U1111-1195-1632 (Registry Identifier: Universal Trial Number)
Record Dates: First submitted 2015-08-31; First posted 2016-02-04 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hematopoietic Stem Cell Transplantation; Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multiple sclerosis autografted patients (Experimental): Individuals with a relapsing-remitting (RRMS) course, secondary progressive (SPMS) or primary progressive (PPMS) were included. Patients should have a Karnofsky performance status (18) above 70% and a EDSS score (1) of 6 or below. The study is approved by the Etichs Committee of the Clinica RUIZ and all patients signed a consent form after being fully informed about procedure an possible complications. Patients included will de treated with Hematopoietic stem cell transplantation
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — autologous transplant using non-frozen peripheral blood stem cells
  Other Names: autologous transplant

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, debilitating disease that causes destruction of central nervous system (CNS) myelin, with varying degrees of axonal damage. It mainly affects young adults and is twice as common in women as in men (1). Studies published from the 1990s brought animal models and theoretical considerations of hematopoietic stem cell transplantation (HSCT) being useful in the prevention and treatment of autoimmune diseases, with clinical responses in some patients, suggesting that high-dose chemotherapy followed by HSCT rescue could "reset" the immunological changes through the control of autoreactive clones, followed by immunological tolerance after immune reconstitution (2); this led to the conclusion that HSCT may be a viable therapeutic option for MS (1-6). Autologous HSCT have been done in patients with MS since 1996 and more than 700 HSCTs have been performed around the world (1-6). Most patients have been treated in small trials or in multicenter studies. In retrospective analyzes, a progression-free survival of more than five years after transplant has been observed, the neurological outcomes being considerably more favorable in patients with the relapsing-remitting type and/or those who showed an inflammatory pattern in magnetic resonance imaging (MRI) during the pre-transplant screening. Reports of good results, particularly in the aggressive forms of MS reinforce the effectiveness HSCT in MS patients with prominent inflammatory activity. The risk of transplant related mortality in HSCT for MS was conventionally considered very high but has declined since 2001 to 1.3% (2-6), this probably being the result of the changes in the conditioning regimens, thus reducing toxicity. Recent data, with more than 700 autologous transplants for MS in Europe, showed an overall survival of 92% in five years and a progression-free survival of 46%, the main cause of mortality and morbidity being the recurrence of the autoimmune disease (2-6). The consensus provides an indication of HSCT in patients with progressive MS unresponsive to conventional therapy and Expanded Disability Status Scale (EDSS) (1) between 3.0 and 6.0. The forms of the disease that might benefit from transplantation are: relapsing remitting, primary or secondary progressive, and the "malignant" form, provided there is evidence of inflammatory activity at the time of transplant indication.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, debilitating disease that causes destruction of central nervous system (CNS) myelin, with varying degrees of axonal damage. It mainly affects young adults and is twice as common in women as in men (1). Studies published from the 1990s brought animal models and theoretical considerations of hematopoietic stem cell transplantation (HSCT) being useful in the prevention and treatment of autoimmune diseases, with clinical responses in some patients, suggesting that high-dose chemotherapy followed by HSCT rescue could "reset" the immunological changes through the control of autoreactive clones, followed by immunological tolerance after immune reconstitution (2); this led to the conclusion that HSCT may be a viable therapeutic option for MS (1-6). Autologous HSCT have been done in patients with MS since 1996 and more than 700 HSCTs have been performed around the world (1-6). Most patients have been treated in small trials or in multicenter studies. In retrospective analyzes, a progression-free survival of more than five years after transplant has been observed, the neurological outcomes being considerably more favorable in patients with the relapsing-remitting type and/or those who showed an inflammatory pattern in magnetic resonance imaging (MRI) during the pre-transplant screening. Reports of good results, particularly in the aggressive forms of MS reinforce the effectiveness HSCT in MS patients with prominent inflammatory activity. The risk of transplant related mortality in HSCT for MS was conventionally considered very high but has declined since 2001 to 1.3% (2-6), this probably being the result of the changes in the conditioning regimens, thus reducing toxicity. Recent data, with more than 700 autologous transplants for MS in Europe, showed an overall survival of 92% in five years and a progression-free survival of 46%, the main cause of mortality and morbidity being the recurrence of the autoimmune disease (2-6). The consensus provides an indication of HSCT in patients with progressive MS unresponsive to conventional therapy and Expanded Disability Status Scale (EDSS) (1) between 3.0 and 6.0. The forms of the disease that might benefit from transplantation are: relapsing remitting, primary or secondary progressive, and the "malignant" form, provided there is evidence of inflammatory activity at the time of transplant indication.

Since 1993 our group has engaged in practicing HSCT using novel methods to both decrease the toxicity of the procedures and diminish costs (7-14); we have done over 400 HSCT for different diseases such as acute leukemia, chronic leukemia, aplastic anemia, myeloma, lymphoma, myelodysplasia and autoimmune diseases, including MS. Within the subset of autologous HSCT, the salient features of our method is that we conduct them on an outpatient basis (8-9, 15-16) and we avoid freezing and thawing the hematopoietic cells in order to both increase viability of hematopoietic cells in the graft and to reduce costs (8-9, 15-16) and we always employ peripheral blood stem cells (PBSC). All these changes have turned the practice of autografting in our hands in an affordable procedure which can be offered to individuals living in underprivileged circumstances such as those prevailing in developing countries (17). Having gained experience autografting hematological malignancies (8-9, 15) we aim to engage in a program of grafting non-cryopreserved autologous hematopoietic stem cells in patients with MS, employing a modification of the autografting conditioning regimen used in malignant diseases.

Material and methods

1. Patients:

   Patients with MS refered to our center for a HSCT will be prospectively entered in the study. Individuals with a relapsing-remitting (RRMS) course, secondary progressive (SPMS) or primary progressive (PPMS). Patients should have a Karnofsky performance status (18) above 70% and a EDSS score (1) of 6 or below. The study has been approved by the Ethics Committee of the Clinic Ruiz and all patients sign a consent form after being fully informed about procedure an possible complications.
2. Peripheral blood stem cell mobilization and apheresis:

   The PBSC mobilization schedule was done with cyclophospha- mide (Cy) and filgrastim (granulocyte colony stimulating factor, G-CSF). Intravenous Cy (50 mg/kg) was delivered in a 120-min period on days -11 and -10. Subcutaneous G-CSF (10 μg/kg/b.i.d.) was delivered on days -9 to -1. Using either a peripheral vein or a Majurkar-type subclavian catheter, the apheresis procedure was performed on day -2, using an Amicus machine (Fresenius Kabi, Deerfield, IL, USA) or a Spectra Optia machine (Terumo BCT, Lakewood, CO, USA) and the Spin-Nebraska protocol [19]. The apheresis objective was to reach at least 1 × 106 viable CD34+ cells/ kg. CD34+ cells in peripheral blood were not measured before the apheresis procedures.
3. Conditioning and autografting:

   As outpatients, intravenous Cy (50 mg(Kg) delivered along a 120 minute period on days -11, -10 , - 2 and - 1 followed by MESNA (1000 mg/m2 along a 180-minute period), ondansetron 8 mg, dexamethasone 4 mg and pantoprazole 40 mg. After the intravenous Cy, ondansetron (4 mg every 12 h after chemotherapy), oral cotrimoxazol (800 / 160 mg every 24 h), oral fluconazole (200 mg) and oral acyclovir (400 mg every 12 h) will be used in all patients until granulocytes were greater than 0.5 x 109/L; in this period all patients will have laboratory workup and clinical studies every 48 h. After the recovery of the granulocytes, patients will be given rituximab (1000 mg total dose along a 3 h period), and in the following six months, cotrimoxazol 800/160 mg bid three times a week, acyclovir 800 mg daily.
4. Apheresis product preservation, studies and infusion:

The products of the apheresis and 1 ml aliquots were kept in ACD-A (Baxter Healthcare, Deerfield IL) at 4oC, in 300 ml transfer packs (Baxter Healthcare, Deerfield IL) composed of gas impermeable, polyvinyl chloride plastic film for up to 72 hours. Enumeration of the total white mononuclear cells (MNC) and CD34 positive cells is done by flow-cytometry (20) in an EPICS Elite ESP apparatus (Coulter Electronics, Hialeah, FL), using for the latter subpopulation the anti-CD34 monoclonal antibody HPCA-2 (Becton Dickinson, San José CA), gating in propidium iodide-excluding CD45(+) MNC population according to forward and 90° angle light scattering. Additional viability studies of the MNC uses propidium iodide exclusion and anti-cell antibodies on a flow cytometer. No purging procedures are performed. The apheresis products obtained on days - 2 and - 1 are reinfused to the patients on days 0 and +1 respectively after keeping them in the conventional blood bank refrigerator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS having a relapsing-remitting course, even though other forms could also qualify: Secondary progressive (SPMS) or primary progressive (PPMS)
* Patients must have a Karnofsky performance status above 70% and a EDSS score of 8 or below.
* In cases of patients with score between 6 and 8 patients will be accepted provided a carer accompanies the patient.
* A recent central nervous system (CNS) MRI study (less than two months).
* Patient has to be able to travel to and remain in Puebla, México during an 4-week period, accompanied by a caregiver.
* Discontinue Immune Modulation or suppression medications 3 months before.

Exclusion criteria:

* EDSS score higher than 8
* Karnofsky performance status lower than 70%
* Been exposed to chemotherapy in the past

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale | 4 years
  EDSS

SECONDARY OUTCOMES:
Overall survival | 4 years
  OS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gale RP, Gomez-Cruz GB, Olivares-Gazca JC, Leon-Pena AA, Gomez-Almaguer D, Gomez-De-Leon A, Gonzalez-Lopez EE, Ruiz-Arguelles A, Soto-Vega E, Munoz-Perez MJ, Ruiz-Delgado GJ, Ruiz-Arguelles GJ. Determine safety of outpatient chemotherapy and autotransplants using refrigerated, non-frozen grafts in persons with multiple sclerosis. Clin Transplant. 2019 Jun;33(6):e13567. doi: 10.1111/ctr.13567. Epub 2019 May 7. PMID 31004516
- [Result] Ruiz-Arguelles GJ, Leon-Pena AA, Leon-Gonzalez M, Nunez-Cortes AK, Olivares-Gazca JC, Murrieta-Alvarez I, Vargas-Espinosa J, Medina-Ceballos E, Cantero-Fortiz Y, Ruiz-Arguelles A, Ruiz-Delgado MA, Ruiz-Delgado RJ, Ruiz-Reyes G, Priesca-Marin M, Torres-Priego MS, Blumenkron-Marroquin D, Ruiz-Delgado GJ. A Feasibility Study of the Full Outpatient Conduction of Hematopoietic Transplants in Persons with Multiple Sclerosis Employing Autologous Non-Cryopreserved Peripheral Blood Stem Cells. Acta Haematol. 2017;137(4):214-219. doi: 10.1159/000469655. Epub 2017 May 18. PMID 28514773
- [Result] Ruiz-Arguelles GJ, Olivares-Gazca JC, Olivares-Gazca M, Leon-Pena AA, Murrieta-Alvarez I, Cantero-Fortiz Y, Gomez-Cruz GB, Ruiz-Arguelles A, Priesca-Marin M, Ruiz-Delgado GJ. Self-reported changes in the expanded disability status scale score in patients with multiple sclerosis after autologous stem cell transplants: real-world data from a single center. Clin Exp Immunol. 2019 Dec;198(3):351-358. doi: 10.1111/cei.13358. Epub 2019 Aug 19. PMID 31394007
- [Derived] Hernandez-Flores EJ, Gallardo-Perez MM, Robles-Nasta M, Montes-Robles MA, Sanchez-Bonilla D, Pastelin-Martinez ML, Ocana-Ramm G, Olivares-Gazca JC, Ruiz-Delgado GJ, Ruiz-Arguelles GJ. Second Autologous Hematopoietic Stem Cell Transplantation in Multiple Sclerosis: A Single-Center Prospective Experience. Transplant Proc. 2024 Jan-Feb;56(1):211-214. doi: 10.1016/j.transproceed.2023.12.004. Epub 2024 Jan 4. PMID 38177042
- [Derived] Montes-Robles MA, Gallardo-Perez MM, Hernandez-Flores EJ, Pastelin-Martinez ML, Sanchez-Bonilla D, Robles-Nasta M, Ocana-Ramm G, Olivares-Gazca JC, Ruiz-Delgado GJ, Ruiz-Arguelles GJ. In persons with CIDP, auto-HSCT can be conducted fully on an outpatient basis and induces significant clinical responses: A prospective study in a single center. Transpl Immunol. 2023 Dec;81:101944. doi: 10.1016/j.trim.2023.101944. Epub 2023 Oct 20. PMID 37866669